CLINICAL TRIAL: NCT01000844
Title: Continuation of Children Enrolled in Protocol #95-011, 'A Randomized Prospective Study for the Prevention of Joint Disease in Children With Severe Factor VIII Deficiency'
Brief Title: Joint Outcome Study Continuation for Children With Severe Factor VIII Deficiency
Acronym: JOSC
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Bayer (Industry); Rush University Medical Center (Other); Phoenix Children's Hospital (Other); The University of Texas Health Science Center, Houston (Other); Oregon Health and Science University (Other); Emory University (Other); University of Texas Southwestern Medical Center (Other); Prisma Health-Midlands (Other); Indiana University School of Medicine (Other); Intermountain Health Care, Inc. (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 01-436
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Hemophilia
Keywords: Hemophilia; Joint; Cartilage; Damage; Prophylaxis; Factor VIII; FVIII; Disease; Arthropathy
MeSH Terms: conditions — Hemophilia A; Disease; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood - EDTA, Citrate Plasma, and DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The original Joint Outcome Study (JOS) enrolled 65 boys with hemophilia from 16 sites nationally. The subjects were randomized to one of two arms (prophylaxis or an enhanced episode-based treatment)and were followed prospectively until the age of six. At the age of six, the proportion of children on each treatment arm who developed bone or cartilage damage as determined by X-Ray or MRI was assessed. In addition, the function and structure of the index joints (defined as knees, ankles, and elbows)were evaluated using a physical assessment scale specially designed for preschool children.

The specific aim of the Joint Outcome Study Continuation (JOSC) is to extend observations of the children participating in the original JOS until the subjects reach the age of 18 years in order to determine the natural history of joint development in hemophilia and the impact of primary or secondary prophylaxis on the prevention, limitation, or reversal of hemophilic arthropathy. In addition, plasma and DNA will be collected and banked yearly for current and future studies of biomarkers and predictors of hemophilia outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the original JOS study, "A Randomized Prospective Study for the Prevention of Joint Disease in Children with Factor VIII Deficiency"
* Written, informed consent of parent or guardian for the proposed study
* The local hemophilia treatment center staff must evaluate the family's participation in the original treatment protocol and determine that the family is capable of complying with the continuation protocol

Exclusion Criteria:

* Unable or unwilling to record the study information

Ages: 8 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study population will be invited based on their enrollment in the original Joint Outcome Study (JOS). This population
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2009-11; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Determine the natuaral history of joint development in hemophilia and the impact of primary or secondary prophylaxis on the prevention, limitation, or reversal of hemophilic arthropathy. | Enrollment, age 14, and study exit at age 18

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Manco-Johnson, MD, Principal Investigator — University of Colorado at Denver Health and Sciences Center

REFERENCES:
- [Derived] Warren BB, Thornhill D, Stein J, Fadell M, Ingram JD, Funk S, Norton KL, Lane HD, Bennett CM, Dunn A, Recht M, Shapiro A, Manco-Johnson MJ. Young adult outcomes of childhood prophylaxis for severe hemophilia A: results of the Joint Outcome Continuation Study. Blood Adv. 2020 Jun 9;4(11):2451-2459. doi: 10.1182/bloodadvances.2019001311. PMID 32492157